CLINICAL TRIAL: NCT02842697
Title: Virtual Hepatic Venous Pressure Gradient (vHVPG) With CT Angiography (CHESS1601): A Prospective Multicenter Study for the Noninvasive Diagnosis of Portal Hypertension
Brief Title: Virtual Hepatic Venous Pressure Gradient (vHVPG) With CT Angiography (CHESS1601)
Acronym: vHVPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing 302 Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, M.D., Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHESS1601
Record Dates: First submitted 2016-07-19; First posted 2016-07-25 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Hypertension, Portal
Keywords: clinically significant portal hypertension; hepatic venous pressure gradient; computed tomographic angiography
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental): Patients will receive CTA, Doppler ultrasound, HVPG measurement, and vHVPG per protocol.
  Intervention: Procedure: HVPG measurement
  Interventions: Procedure: HVPG measurement; Procedure: CTA; Procedure: Doppler ultrasound

INTERVENTIONS:
Procedure: HVPG measurement — HVPG obtained by means of catheterization of a hepatic vein with a balloon catheter
Procedure: CTA — Three-dimensional hepatic vein-portal vein model constructed with CTA images
Procedure: Doppler ultrasound — Portal vein velocity measured by Doppler ultrasound

SUMMARY:
This is a prospective, multi-center trial conducted at 1 Guangzhou and 2 Beijing centers designed to determine the diagnostic performance of virtual hepatic venous pressure gradient (vHVPG) (investigational technology) by anatomic computed tomographic angiography (CTA) for non-invasive assessment of the clinically significant portal hypertension (CSPH) in patients with compensated cirrhosis. Direct hepatic venous pressure gradient (HVPG) measurement by means of catheterization of a hepatic vein with a balloon catheter is the gold-standard method to assess the presence of CSPH, which is defined as HVPG≥10 mmHg.

DETAILED DESCRIPTION:
This is a prospective, multi-center trial conducted at 1 Guangzhou (Nanfang Hospital) and 2 Beijing (Beijing 302 Hospital, Beijing Shijitan Hospital) centers designed to determine the diagnostic performance of vHVPG (investigational technology) by anatomic CTA for non-invasive assessment of the CSPH in patients with compensated cirrhosis. Direct HVPG measurement by means of catheterization of a hepatic vein with a balloon catheter is the gold-standard method to assess the presence of CSPH, which is defined as HVPG≥10 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients providing written informed consent
* Patients with compensated cirrhosis and scheduled to undergo clinically-indicated invasive HVPG measurement by means of catheterization of a hepatic vein with a balloon catheter
* Has undergone > 64 multi-detector row CTA within 14 days prior to hepatic vein catheterization
* No hepatic-portal vein interventional therapy between the CTA and hepatic vein catheterization

Exclusion Criteria:

* Prior transjugular intrahepatic portosystem stent-shunt surgery
* Prior devascularization operation
* Has received a liver transplant
* Patients with known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status
* Patient requires an emergent procedure
* Any active, serious, life-threatening disease
* Inability to adhere to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of vHVPG | 1 day
  Diagnostic accuracy of vHVPG to determine presence or absence of a CSPH when compared to HVPG as the reference standard (HVPG≥10mmHg)

SECONDARY OUTCOMES:
Diagnostic Performance of vHVPG | 1 day
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of vHVPG when compared to HVPG as the reference standard (HVPG≥10mmHg)
vHVPG Numerical Correlation | 1 day
  Correlation of the vHVPG numerical value with the HVPG numerical value

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (3):
- China (3):
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] de Franchis R, Dell'Era A. Invasive and noninvasive methods to diagnose portal hypertension and esophageal varices. Clin Liver Dis. 2014 May;18(2):293-302. doi: 10.1016/j.cld.2013.12.002. Epub 2014 Feb 25. PMID 24679495
- [Background] Berzigotti A, Seijo S, Reverter E, Bosch J. Assessing portal hypertension in liver diseases. Expert Rev Gastroenterol Hepatol. 2013 Feb;7(2):141-55. doi: 10.1586/egh.12.83. PMID 23363263
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Qi X, Li Z, Huang J, Zhu Y, Liu H, Zhou F, Liu C, Xiao C, Dong J, Zhao Y, Xu M, Xing S, Xu W, Yang C. Virtual portal pressure gradient from anatomic CT angiography. Gut. 2015 Jun;64(6):1004-5. doi: 10.1136/gutjnl-2014-308543. Epub 2014 Nov 14. No abstract available. PMID 25398771
- [Result] Qi X, An W, Liu F, Qi R, Wang L, Liu Y, Liu C, Xiang Y, Hui J, Liu Z, Qi X, Liu C, Peng B, Ding H, Yang Y, He X, Hou J, Tian J, Li Z. Virtual Hepatic Venous Pressure Gradient with CT Angiography (CHESS 1601): A Prospective Multicenter Study for the Noninvasive Diagnosis of Portal Hypertension. Radiology. 2019 Feb;290(2):370-377. doi: 10.1148/radiol.2018180425. Epub 2018 Nov 20. PMID 30457484